CLINICAL TRIAL: NCT03601650
Title: The Effect of Mindful Eating on Calorie Intake and Diet Over a 3-day Period Among Healthy Weight Women.
Brief Title: The Effect of Mindful Eating on Calorie Intake and Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Responsible Party: Principal Investigator, Katy Tapper, Dr Katy Tapper, City, University of London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSYETH (R/L) 16/17 92
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Diet Modification
MeSH Terms: interventions — Eating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindful eating (Experimental): Participants will be encouraged to focus on the sensory properties of their food every time they eat. This will be achieved via an audio recording that they will listen to in the laboratory at their first appointment and that they will have access to over the three-day intervention period. They will also receive a pack of envelopes to open over the intervention period that will also contain reminders to focus on the sensory properties of their food every time they eat.
  Interventions: Behavioral: Mindful eating
- Eating without distractions (Active Comparator): Participants will be encouraged to eat their food without distractions every time they eat. This will be achieved via an audio recording that they will listen to in the laboratory at their first appointment and that they will have access to over the three-day intervention period. They will also receive a pack of envelopes to open over the intervention period that will also contain reminders to eat their food without distractions every time they eat.
  Interventions: Behavioral: Eating without distractions
- No strategy control (No Intervention): Participants will simply complete the measures

INTERVENTIONS:
Behavioral: Mindful eating — Attending to the sensory properties of food as it is eaten
  Other Names: Attentive eating
  Arms: Mindful eating
Behavioral: Eating without distractions — Eating without intentionally attending to something else such as a television, smartphone, computer, book etc
  Arms: Eating without distractions

SUMMARY:
The study will examine the effect of focussing on the sensory properties of food whilst eating. It will look at effects on calorie intake and diet over a 3-day period among women of a healthy weight. Participants asked to focus on the sensory properties of their food will be compared with a second group of participants who will be asked to eat their food without distractions and a third group who will not be provided with any strategy.

DETAILED DESCRIPTION:
The research will be conducted as a between subject design over a period of three days (Tuesday-Thursday). Upon arrival at the laboratory (on a Monday), participants will be provided with more information about the study and will complete a demographics questionnaire. A smartphone app will be downloaded onto the participant's phone and the participant will be provided with login details to access the food diary Intake24. Participants will be asked to complete the food diary every night over a period of three days. The diary will ask participants to record what they consumed for breakfast, lunch, dinner, as well as snack on a daily basis. All participants will receive a reminder notification on their phone each evening during the 3-day period to complete the Intake 24 food diary. They will also be asked to rate how well they think they remembered the food they had eaten that day.

During the 3-day period, some participants will also be asked to open reminders in sealed envelopes at particular times of the day. The app will additionally include a recording that participants will be able to listen to at their own convenience, as many times as they wish.

The content of the reminders and recording will differ between participants depending on the condition they are allocated to. There will be three conditions: intervention, no distraction control, and no strategy control.

In the intervention condition, participants will open reminders related to focusing on the sensory properties of their food while eating their meals. These participants will also have access to a recording that will encourage them to focus on the sensory properties of the food (e.g. its smell, look, texture).

Participants in the no distraction control condition will open reminders related to eating their meals with no distractions. The recording provided to participants in this condition will encourage them to consume their meals with no surrounding distractions (e.g. to avoid watching television or listening to the radio). During the study, the number of times the recording is played as well as the date and time it is played will be recorded.

In the intervention and no distraction control group, at the end of each of the three days participants will also be asked to rate the extent to which they adhered to the strategy they were provided with.

In the no strategy control condition, participants will not receive any reminders to open or have access to a recording.

After the three days (i.e. on a Friday), participants will return to the laboratory. They will be asked to complete a questionnaire regarding the usability of the mobile app and the online food diary. Via this questionnaire, they will also be asked about whether they thought taking part in the study influenced their eating behaviour and the amount of pleasure they got from their food during the three-day period. Additionally they will complete a questionnaire measuring sensitivity to reward. At this session participants will be asked if they are happy to have their weight and height measured. If they are, the researcher will measure their weight and height.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speaker
* BMI of 20 to 25 based on reported weight and height
* Access to data or wifi during the evenings

Exclusion Criteria:

* Dieting to lose weight
* Taking medication that may affect appetite
* Current or previous diagnosis of an eating disorder
* Completion of related studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Calorie intake | Three days during intervention delivery
  Total calorie intake over three days

SECONDARY OUTCOMES:
Intake of non milk extrinsic sugars | Three days during intervention delivery
  Total intake (in grams) of non milk extrinsic sugars over the three days
Intake of saturated fat | Three days during intervention delivery
  Total intake (in grams) of saturated fat over the three days
Fruit and vegetable intake | Three days during intervention delivery
  Total intake (in grams) of fruit and vegetables, excluding juices, smoothies, potatoes and legumes
Intake of fibre | Three days during intervention delivery
  Total intake (in grams) of fibre (using the Englyst measure)

CONTACTS AND LOCATIONS:
Overall Officials: Katy Tapper, PhD, Principal Investigator — City, University of London
Locations (1):
- City, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No